CLINICAL TRIAL: NCT03753828
Title: Estimated Impact of Fungal Colonization in Cystic Fibrosis From Secondary Exploitation of MucoFong Database.
Acronym: MucoFong2
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2017/34
Record Dates: First submitted 2018-09-12; First posted 2018-11-27 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2018-08

CONDITIONS: Cystic Fibrosis Lung
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Cystic Fibrosis sputum mycological analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients de novo colonized by fungi: Patients in Cystic Fibrosis de novo colonized by fungi during their follow-up

SUMMARY:
The main objective of the project "MucoFong" (19021906 national french program n which Vaincre La Mucoviscidose participated: N82006/ 351) was to determine the fungi present the respiratory tract of CF patients responsible for either colonization or authentic infectious diseases. The Mucofong data allowed the team to provide for the 1st time national French guidelines for the management of CF sputum mycological analysis (MucoMicrobes work group coordinated by Prof. Plésiat published in 2015 in the REMIC book). Nevertheless, the team has a comprehensive database that it still has to analyze beyond these initial results. The main goal today is to clarify the role of fungi in the lung function degradation of these patients by studying the overall risk and estimated impact of fungal colonization in our cohort.

DETAILED DESCRIPTION:
The material includes data from the followup of the 300 patients (3 visits per patient for which the team collected and verified the biological radiological and clinical data).

Relations between Aspergillus fumigatus or Candida albicans and lung function or clinical outcome of patients will be longitudinally analyzed taking as output variable FEV1, according to bibliography data available.

To assess the attributed fungal risk, the team will focus on the 57 patients de novo colonized by fungi at the second visit. Three physician experts will determine the impact of such fungal colonization on the patient clinical and respiratory parameters.

The expert conclusion concordance and statistical significance will be evaluated using the kappa score.

This project will be realized in collaboration with the groups of Prof. R. Thiebaut (Methodology and Epidemiology Service Bordeaux University Hospital, INSERM U1219 / INRIA SISTM) and Prof. M. Fayon (Department of Pediatrics, Pediatric reference centre) University Hospital of Bordeaux.

ELIGIBILITY:
Inclusion Criteria:

All patients included in the database meet the following criteria:

* Patient whose diagnosis of cystic fibrosis has been validated on the criteria in force,
* Patient usually followed in one of the 7 centers involved in the PHRC,
* Patient aged at least 6 years without an upper age limit,
* Patient benefiting from a mycological assessment carried out in the context of the usual microbiological monitoring (good clinical practice),
* Cystic fibrosis Patient benefiting from a mycological assessment carried out in front of a clinical episode of aggravation requiring biological exploration,
* Patient who has signed informed consent at the time of inclusion,-patient affiliated with a social security scheme.

Exclusion Criteria:

Patients meeting the following criteria were not included in the database:

* Pulmonary transplant Patient,
* Patient or their parents (if the patient is a minor) refusing any participation in the study,
* Major incapable subject, under guardianship or under the protection of Justice,
* Refusal or inability to give informed consent.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 300 patients followed for 2 years including a subpopulation of 40 patients with pro-and eukaryotic respiratory microbiota documented by high-throughput sequencing.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2018-10-13 (Actual); Study Completion 2018-10-13 (Actual)

PRIMARY OUTCOMES:
Describe the micromycetes find in lung in patients with cystic fibrosis | Day 1
  Relation between the micromycetes and the pathologic lung in patients with cystic fibrosis

SECONDARY OUTCOMES:
Number of patient with a. fumigatus, c. albicans or other micromycete | Day 1
  Establish the proportion of patients of a colonization in a. fumigatus, in c. albicans or other micromycete, carriers from awareness of a. fumigatus (unlike an ABPA)
Detect, from data of high-throughput sequencing, combinations of bacteria or fungi are present and clear profile of affinity between genres, in patients with cystic fibrosis. | Day 1
  Detect, from data of high-throughput sequencing, combinations of bacteria or fungi are present and clear profile of affinity between genres, in patients with cystic fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Laurence DELHAES, MD/PhD, Principal Investigator — Hospital University, Bordeaux
Locations (1):
- University Hospital, Bordeaux, Bourdeaux, France